CLINICAL TRIAL: NCT01761513
Title: A Randomized,Open Label,Active-controlled, Multiple Dosing and Crossover Clinical Trial to Evaluate the Safety and Pharmacokinetics/Pharmacodynamics of YH4808 After Postprandial Oral Administration in Healthy Volunteers
Brief Title: YH4808 Postprandial PK/PD Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH4808-107
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — YH4808; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental)
  Interventions: Drug: YH4808
- Sequence 2 (Experimental)
  Interventions: Drug: YH4808
- Sequence 3 (Active Comparator)
  Interventions: Drug: YH4808
- Sequence 4 (Active Comparator)
  Interventions: Drug: YH4808

INTERVENTIONS:
Drug: YH4808 — Group1
  1. adminitration of YH4808 dose1, bid for 2weeks
  2. wash-out period for 3weeks between period1 and period2
  3. adminitration of YH4808 dose2, qd for 2weeks
Drug: YH4808 — Group2
  1. adminitration of YH4808 dose2, qd for 2weeks
  2. wash-out period for 3weeks between period1 and period2
  3. adminitration of YH4808 dose1, bid for 2weeks
Drug: YH4808 — Group3
  1. adminitration of YH4808 dose2, bid for 2weeks
  2. wash-out period for 3weeks between period1 and period2
  3. adminitration of Nexium tab 40mg, bid for 2weeks
  Other Names: YH4808, Nexium
Drug: YH4808 — Group 4
  1. adminitration of Nexium tab 40mg, bid for 2weeks
  2. wash-out period for 3weeks between period1 and period2
  3. adminitration of YH4808 dose2, bid for 2weeks
  Other Names: Nexium

SUMMARY:
A clinical Study to evaluate the safety and pharmacokinetics/pharmacodynamics(PK/PD) of YH4808 after repeated Oral administration and Postprandial state in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged 20 to 55 with a body mass index(BMI) between 18.5 and 25 kg/m2
2. Subject who has no congenital, chronic diseases and disease symptoms in medical examination result
3. Subject who shows negative reaction of UBT(Urea Breath Test)
4. Subject who is judged to be eligible by principal investigator or sub-investigator according to various reasons including their abnormal test results (clinical laboratory test, chest X-ray test, 12-lead ECG etc) 4 weeks before the first IP adminitration
5. Medically acceptable contraception(including individuals who are medically unable to become pregnant) used during the clinical trial
6. Volunteers who has signed a written informed consent voluntarily, prior to any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the purpose, contents, and characteristic of the drug

Exclusion Criteria:

1. Subject who is hypersensitive to components contained in YH4808 or this drug
2. Subject who has history or presence of clinically significant diseases in liver, kidney, gastrointestinal tract, nervous system, respiratory system, endocrine system, blood tumor, cardiovascular, urinary system, and mental disorder
3. Subject who has history of surgical operation or diseases related to gastrointestinal symtem (e.g. crohn's disaese, ulcer etc except appendectomy or simple for herina)
4. Other exclusions apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve of YH4808 | Blood sampling during 0 ~ 24 hrs after administration
Peak plasma concentration of YH4808 | Blood sampling during 0~24 hrs after administration

SECONDARY OUTCOMES:
Time to reach peak plasma concentration of YH4808 | Blood sampling during 0 ~ 24 hrs after administration

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, Ph.D, M.D., Principal Investigator — Yonsei University Health System(Severance Hospital)
Locations (1):
- Yonsei University Health System(Severance Hospital), Seoul, Seodaemun-gu,Sinchon-dong, South Korea

REFERENCES:
- [Derived] Yoon S, Oh E, Park MS, Jang SB, Byun HM, Park H, Kim H, Kim CO. Comparison of the pharmacokinetics and pharmacodynamics of YH4808 in healthy subjects for defining an appropriate dosing regimen. Transl Clin Pharmacol. 2021 Sep;29(3):150-159. doi: 10.12793/tcp.2021.29.e15. Epub 2021 Sep 17. PMID 34621707